CLINICAL TRIAL: NCT03854110
Title: Phase 1 Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of GP-2250 With Gemcitabine in Advanced Unresectable or Metastatic Pancreatic Adenocarcinoma Following Progression on 5-FU-based Chemotherapy
Brief Title: Trial to Evaluate Safety and Tolerability of GP-2250 in Combination With Gemcitabine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP-2250-1001
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer, Adult
Keywords: Advanced disease; 5-fluorouracil
MeSH Terms: conditions — Pancreatic cancer, adult | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GP-2250 Monotherapy (Experimental): GP-2250 in doses of 250 mg up to 30 grams intravenously on Days -7, 1, 8, 15 (Cycle 1) and Cycle 2 and all subsequent cycles on Days 7, 8, 15 of a 28-day cycle with gemcitabine 1000 mg/m2 on Days 1, 8, 15 days of the cycle.
  Interventions: Drug: GP-2250

INTERVENTIONS:
Drug: GP-2250 — GP-2250 monotherapy for pharmacokinetics and safety; GP-2250 plus gemcitabine for safety, tolerability, pharmacokinetics, and biomarker assessments
  Other Names: gemcitabine

SUMMARY:
This is a phase 1 first in human, dose escalation trial of GP-2250 administered in combination with gemcitabine in subjects with advanced pancreatic cancer previously treated with 5-fluorouracil-based chemotherapy.

Prior radiosensitization with gemcitabine, the use of 5-fluorouracil, FOLFIRINOX or Nab-paclitaxel/gemcitabine in the neoadjuvant setting, and prior pancreaticoduodenectomy (Whipple procedure) is allowed. If prior treatment with gemcitabine was at therapeutic doses, a minimum of 3 months must have elapsed since the end of such treatment.

As a precursor to 5-FU use of capecitabine-based chemotherapy is also permitted.

DETAILED DESCRIPTION:
This trial used a Bayesian Optimal Interval (BOIN) dose escalation design of GP-2250 as a single-dose monotherapy (Cycle 1 only) followed by combination therapy with gemcitabine for Cohorts 1 through 5. Following implementation of Amendment 7 and beginning with dose Cohort 6 and all subsequent cohorts, the trial will use a 3+3 dose escalation design, and will continue as single-dose monotherapy (Cycle 1 only) followed by combination therapy with gemcitabine. Subjects will continue to receive treatment until disease progression assessed by RECIST V1.1 criteria, clinical disease progression as assessed by the Investigator, development of a dose limiting toxicity, unacceptable toxicity, subject request for withdrawal, Investigator assessment that risk outweighs benefit, or study closure by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent:

1. Capable of giving signed informed consent as described in Appendix 1: Regulatory, Ethical, and Trial Oversight Considerations which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Male and female subjects age > 18 years at the time of trial entry. Type of Subject and Disease Characteristics
3. Histologically or cytologically confirmed advanced unresectable or metastatic pancreatic adenocarcinoma
4. Subjects should be eligible to receive gemcitabine monotherapy for the treatment of their pancreatic cancer per the judgment of the Investigator
5. Subjects must have documented disease progression while receiving or within 3 months of completing prior treatment with 5-fluorouracil-based chemotherapy.
6. Subjects must have at least one RECIST Version 1.1 defined measurable tumor lesion
7. Subjects must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1.
8. Subjects with known central nervous system metastasis must have undergone brain targeted treatment and must be asymptomatic or radiographically and clinically stable (including not requiring steroids or anti-seizure medications) for at least 4 weeks prior to enrollment.
9. All subjects must consent to provide archived tumor specimens for biomarker studies.
10. Subjects must have adequate organ function as indicated by the following laboratory values:

    1. Absolute neutrophil count (ANC) ≥ 1,500 /mL
    2. Platelets ≥ 100,000 / mL
    3. Hemoglobin ≥ 9 g/dL
    4. Serum creatinine ≤ 1.5 X upper limit of normal (ULN)
    5. Serum total bilirubin ≤ 1.5 × ULN
    6. Aspartate aminotransferase (AST), (Serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT), and (Serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 × ULN OR ≤ 5 × ULN for subjects with liver metastasis
    7. International Normalized Ratio (INR) and/or Prothrombin Time (PT) ≤ 1.5 × ULN
    8. Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN
    9. Serum Albumin ≥ 3 gm/dL
11. Female subjects of childbearing potential (woman of childbearing potential [WOCBP]) must have a negative serum pregnancy test.
12. Subjects must use adequate contraception for the duration of the trial:

    1. Male subjects must agree to use a highly effective contraception during the treatment period and for at least 3 months after the last dose of trial intervention and refrain from donating sperm during this period
    2. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a WOCBP OR a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of trial intervention.

Exclusion Criteria:

1. Diagnosis of any active malignancy other than pancreatic cancer within the past 2 years (not including non-melanoma skin carcinoma, ductal carcinoma in situ of the breast, or carcinoma in situ of uterine cervix treated with curative intent).
2. Subjects has a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonia or multiple allergies, clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome with <=6 months prior to the start of study treatment, symptomatic or uncontrolled arrhythmia, congestive heart failure, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or ascites requiring paracentesis in the 4 weeks prior to Screening.
3. Any other medical, psychiatric, or social condition deemed by the Investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate and participate in the trial, or which would interfere with the interpretation of the results.
4. Subject has undergone major surgery, other than diagnostic surgery (ie, surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
5. Prior history or current signs of hyphema or glaucoma.
6. History of sickle cell disease or hereditary non-spherocytic hemolytic anemia.
7. Baseline QTc interval >480 msec for female subjects or >450 msec for male subjects.
8. Subject is unwilling or unable to comply with study procedures or is planning to take a vacation for 7 or more consecutive days during the source of the study.
9. First degree relative of the investigator, study staff or the sponsor.
10. Positive test for SARS-CoV2 (COVID-19) by polymerase chain reaction (PCR) testing within one week prior to Screening.
11. Any chemotherapy administered within 3 weeks or 5 half-lives (whichever is shorter) before first dose of GP-2250; other anti-cancer therapy (including surgery, radiotherapy, immunotherapy, hormone therapy, or targeted therapy) administered within 4 weeks or 5 half-lives (whichever is shorter) before the first dose of GP-2250; or within 6 weeks in the case of certain therapies (mitomycin C and nitrosoureas).

    Prior/Concurrent Clinical Trial Experience:
12. Investigational therapy administered within 4 weeks or 5-half lives (whichever is shorter) before the first dose of GP-2250.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 12-24 months
  Dose Limiting Toxicity - dose at which toxicity causes cessation of dose escalations.

SECONDARY OUTCOMES:
Carbohydrate Antigen 19-9 (CA-19-9) | 12-24 months
  A type of antigen released by pancreatic cancer cells and usually changes as disease progression or regressions occurs. Measurement of changes, if any, will be assessed in each patient.
Effect on disease | 6-12 months
  To assess the preliminary efficacy of GP 2250 in combination with gemcitabine

CONTACTS AND LOCATIONS:
Overall Officials: Anup Kasi, MD, Study Chair — University of Kansas
Locations (5):
- United States (5):
  - Hoag Family Cancer Institute, Newport Beach, California
  - University of Kansas Cancer Center, Fairway, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Abramson Cancer Center at the University of Pennsylvania, Phildelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchholz M, Majchrzak-Stiller B, Hahn S, Vangala D, Pfirrmann RW, Uhl W, Braumann C, Chromik AM. Innovative substance 2250 as a highly promising anti-neoplastic agent in malignant pancreatic carcinoma - in vitro and in vivo. BMC Cancer. 2017 Mar 24;17(1):216. doi: 10.1186/s12885-017-3204-x. PMID 28340556
- [Background] Majchrzak-Stiller B, Buchholz M, Peters I, Waschestjuk D, Strotmann J, Hohn P, Hahn S, Braumann C, Uhl W, Muller T, Mohler H. GP-2250, a novel anticancer agent, inhibits the energy metabolism, activates AMP-Kinase and impairs the NF-kB pathway in pancreatic cancer cells. J Cell Mol Med. 2023 Jul;27(14):2082-2092. doi: 10.1111/jcmm.17825. Epub 2023 Jun 30. PMID 37390227
- [Background] Kim MS, Glassman D, Handley KF, Lankenau Ahumada A, Jennings NB, Bayraktar E, Foster K, Joseph R, Lee S, Coleman RL, Sood AK. Mechanism and rational combinations with GP-2250, a novel oxathiazine derivative, in ovarian cancer. Cancer Med. 2024 Aug;13(15):e70031. doi: 10.1002/cam4.70031. PMID 39114948